CLINICAL TRIAL: NCT06130644
Title: Early Lymph Node Metastasis in T1/2 Stage Colorectal Cancer: Molecular and Clinical Insights
Status: Completed | Type: Observational
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: PRSYM202311
Record Dates: First submitted 2023-11-01; First posted 2023-11-14 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with lymph node metastasis: T1/2N+ patients
- Patients without lymph node metastasis: T1/2N- patients

SUMMARY:
The prognostic implications of lymph node metastasis in colorectal cancer patients at an early stage, specifically T1/2 stage, are relatively unfavorable. Therefore, understanding the clinical and molecular traits relevant to metastasis in T1/2 stage are of substantial clinical importance.

DETAILED DESCRIPTION:
Patients were classified based on their lymph node staging, with an ancillary categorization into MSI-H and MSS subgroups. A comparative mutational study was performed among these groups, incorporating risk stratification and Receiver Operating Characteristic curve analysis, with the aim of discerning the predictability of clinical features integrated with molecular characteristics for early metastasis in T1/2 stage colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18-75 years old;
* Clinical staged T2;
* Histologically proven colon or rectal adenocarcinoma.

Exclusion Criteria:

* Patients over 80 years of age;
* Recurrent colorectal cancer;
* Multiple primary tumors;
* Distant metastasis.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Colorectal cancer patients.
Sampling Method: Non-Probability Sample
Enrollment: 1451 (Actual)
Dates: Start 2003-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
MSI status | through study completion, an average of 1 year
  (I) MSI-High (MSI-H) if two or more mononucleotide markers in tumor tissue had size variations of ≥3bp compared to normal tissue; (II) MSI-Low (MSI-L) if a single mononucleotide marker in tumor tissue exhibited a size variation of ≥3bp compared to normal tissue; (III) Microsatellite Stable (MSS) if there were no size variations of ≥3bp in mononucleotide markers in tumor tissue compared to normal tissue.

SECONDARY OUTCOMES:
Somatic Mutation Distribution | through study completion, an average of 1 year
  targeted NGS
Tumor Mutation Burden (TMB) | through study completion, an average of 1 year
  targeted NGS

IPD SHARING:
Plan to Share IPD: No